CLINICAL TRIAL: NCT05905575
Title: A Family Dyad-focused Diabetes Self-Management Intervention for African American Adults With Type 2 Diabetes
Brief Title: A Family Dyad-focused Diabetes Self-Management Intervention for African American Adults
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Ohio State University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2023 H0010
Record Dates: First submitted 2023-04-18; First posted 2023-06-15 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Intervention Model Description: This two-arm randomized controlled trial (RCT) will test the feasibility, acceptability and efficacy of a family-dyad-focused intervention. A convenience sample will be recruited at clinics/pharmacy at Central Ohio. We will enroll a total of 208 participants in the study with104 African-Americans with T2D and one family member of each patient (104 patient-family member dyads). Patients with T2D will be randomized 1:1 to the intervention or control arm (n=52/arm). The family member of each patient will receive the same treatment as that assigned to the patient.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Patient-family member dyads in the family dyad intervention arm will receive 1) 10 sessions (8 weekly and 2 biweekly) over 12 weeks of family-dyad-focused, virtual group sessions on diabetes self-management and family support; 2) family dyad-focused support component in each group session; and 3) individual family feedback telephone sessions.
  Interventions: Behavioral: Family dyad diabetes intervention
- Control (No Intervention): All control participants will receive usual care from their primary healthcare provider. A condensed family dyad diabetes intervention will be delivered to the control participants by the end of the study.

INTERVENTIONS:
Behavioral: Family dyad diabetes intervention — The goals of the intervention are to encourage participants to (1) daily self-manage diabetes and stress; (2) establish a healthy eating pattern; (3) engage in brisk walking of 150 or more minutes a week; and (4) use solution-focused problem-solving strategy and supportive family communication skills.
  Arms: Intervention

SUMMARY:
A family dyad-focused diabetes self-management for African American adults with type 2 diabetes is a randomized controlled trial (RCT) that aims to test the feasibility, acceptability, and efficacy of a family-dyad focused intervention on glycemic control (hemoglobin A1c) and health-related quality of life (HRQOL) in African American adults with type 2 diabetes (T2D).

DETAILED DESCRIPTION:
Eligible participants and their family members will be randomly assigned to either the intervention and control group. Patient-family-member dyads in the intervention arm will virtually receive 1) 10 session over 12 weeks of family dyad-focused, group sessions on diabetes self-management and family support; 2) family dyad-focused support component in each group session; and 3) individual family feedback telephone sessions. All participants will be assessed at baseline, post-intervention and six months after intervention.

ELIGIBILITY:
Inclusion Criteria:

Individual with type 2 diabetes:

* Self-identification as African American;
* 40 years or older
* Type 2 diabetes diagnosis for at least six months;
* A1c > 7.0% at time of enrollment;
* Being able to speak and read English;
* Being able to walk;
* Having an adult family member/close friend willing to co-participate in the study.

Family members:

* Adults (18 years or older, with or without T2D);
* Residing in the same household as the T2D participants;
* Being a spouse, adult child or sibling; or close friend
* Being able to walk;
* Being able to speak and read English.

Exclusion Criteria:

Individual with T2D and family members:

* Being pregnant or have an advanced or terminal condition;
* Being cognitively impaired or unable to provide informed consent;
* Lack conclusive evidence of T2D for patients with T2D.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 208 (Estimated)
Dates: Start 2023-06-01 (Actual); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
Change in diabetes control | Baseline (T1) to immediate post-intervention at month 5 (T2)
  Change in glycosylated hemoglobin A1c will be measured with finger stick blood with a glycosylated hemoglobin A1CNow+ test. Changes in average percent of A1c will be used in the study.
Change in diabetes control | Baseline (T1) to six months after intervention (T3) at month 11
  Change in glycosylated hemoglobin A1c will be measured with finger stick blood with a glycosylated hemoglobin A1CNow+ test. Changes in average percent of A1c will be used in the study.
Change in health-related quality of life | Baseline (T1) to immediate post-intervention at month 5 (T2)
  Patient-Reported Outcomes Measurement Information System Global Health (PROMIS 10) will be used to measure changes in total scores of the global physical and global mental health. Scores range from 0-100 with higher scores indicating better quality of life.
Change in health-related quality of life | Baseline (T1) to six months after intervention (T3) at month 11
  Patient-Reported Outcomes Measurement Information System Global Health (PROMIS 10) will be used to measure changes in total scores of the global physical and global mental health. Scores range from 0-100 with higher scores indicating better quality of life.

SECONDARY OUTCOMES:
Change in blood pressure control | Baseline (T1) to immediate post-intervention at month 5 (T2)
  Change in blood pressure will be measured with average scores of systolic and diastolic pressures.
Change in blood pressure control | Baseline (T1) to six months after intervention (T3) at month 11
  Change in blood pressure will be measured with average scores of systolic and diastolic pressures.

CONTACTS AND LOCATIONS:
Locations (1):
- The Ohio State University College of Nursing, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: Yes
Data will be made available to the public as immediately and broadly as possible while safeguarding the privacy of participants and protecting confidential and proprietary data. All research data will be shared as requested in accordance with federal regulations, the Freedom of Information Act (FOIA). Requests from researchers will be reviewed by the project investigators, and we will provide the requesting researcher with the minimum necessary data; the shared data will not have any individual participant identifiers or specific clinic identifiers.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be made available to the public as immediately and broadly as possible while safeguarding the privacy of participants and protecting confidential and proprietary data.
Access Criteria: Requests will be reviewed by the project investigators (PI). In accordance with NIH policies and procedures regarding data use and data sharing, user registration will be required to access the les. Users must agree to the conditions of use governing access to the public release data, including restrictions against attempting to identify study participants, destruction of the data after analyses are completed, reporting responsibilities, restrictions on redistributions of the data to third parties, and proper acknowledgement of the data resource. Any presentations, abstracts, or publications must include an acknowledgement/reference of the research team.
  The requesting researcher(s) will be notified that they may only use the data for the purposes for which the data were requested and only by the individuals listed in the request. The requesting researcher(s) will be responsible for notifying the PI upon completion of analysis indicating the way the data were destroyed.

REFERENCES:
- [Derived] Hu J, Mion LC, Tan A, Bartle-Haring S, Miller C, Joseph JJ. Family dyad-focused diabetes self-management intervention (FDSMI) for African American adults with type 2 diabetes: Study protocol. Contemp Clin Trials. 2025 Sep;156:108029. doi: 10.1016/j.cct.2025.108029. Epub 2025 Jul 22. PMID 40706841